CLINICAL TRIAL: NCT02024802
Title: Clinical Trial: Transdermal Compounded Pain Creams and Patient Pain Perception
Brief Title: Compounded Pain Creams and Patient Perception
Status: Withdrawn | Type: Observational
Sponsor: Marwood LowCost Pharmacy (Other)
Responsible Party: Sponsor
Other Study IDs: MLP-001-PC
Record Dates: First submitted 2013-12-28; First posted 2013-12-31 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Neurologic Pain; Nociceptive Pain
Keywords: Pain; Pain Cream; Nociceptive pain; neurologic pain; transdermal; compounding; compound
MeSH Terms: conditions — Nociceptive Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There has been a significant increase in the number of prescriptions being filled for Custom Compounded Pain Creams. This study serves to evaluate the patient perception and satisfaction with this type of pain therapy allowing us to identify any statistically relevant relationships that may exist between this type of therapy and patient pain perception. A secondary goal would be to identify any significantly relevant relationships that may exist between this change in pain perception (if any) and the patients overall sense of well-being. The investigators' null hypothesis is that greater that 85% of people will see an significant decrease in perceived pain levels and greater than 85% increase in patient overall sense of well being.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the level of pain perceived by chronic neuropathic and/or inflammatory pain patients using a compounded transdermal pain cream as a pain management solution. Our goal is to identify statistically relevant relationships existing between this type of pain therapy and patients' perceived pain levels.

A secondary goal of this study is to identify any statistically relevant relationships between this change in pain perception (if any) and the patient's perception of overall well-being.

This will be an observational study with a cohort observational model study design. Patients whom have been prescribed a compounded pain cream regimen as a new pain therapy but have not yet begun the regimen will be recruited.

We will work with local prescribing neurologic, orthopedic and pain clinic physicians to identify patients who will be beginning this type of therapy in the near future. Prior to administering their first dose, the participants will need to complete the consenting process. Participants may opt to review and complete the informed consent form with their doctor or with a member of the pharmacy research team.

The custom survey entitled MLP-001-PC will be administered throughout the 12 week study at 4 week intervals (baseline, 4 weeks, 8 weeks, and 12 weeks).

Participants will not be required to come to the pharmacy to complete the subsequent surveys. They can be mailed or emailed at the participant's discretion. Any patient whom opts to receive their survey via mail or email will need to indicate so on their patient information form and provide a signature at that time stating that all surveys will be completed on one's own behalf (See Attachment 1).

If the participants opt to receive their surveys by mail, we will ask that they return their survey to the pharmacy either in person or in the stamped envelope that will be provided. Participants receiving their surveys by email, will need to return their completed surveys in person, by mail or by email.

We will follow up with the patients at 3 and 6 days after the distribution of the surveys to remind them to complete and return the surveys. Surveys which are not completed within one week of the respective follow-up date will be excluded from the study for that respective follow-up interval. These participants will still be encouraged to complete the next survey for the next follow-up date.

The study is projected to last one year from enrollment of the first subject to completion of the last subject's participation.

All results from the baseline and follow-up surveys will be scored and the data will be compiled on site. Statistical analysis (Multinomial Regressional Analysis) will be performed to identify all statistically relevant correlations. All data will be summarized and concluded.

A description of this clinical trial will be available on http://ClinicalTrials.gov, as required by U.S. Law.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be in the range of 18 to 85 years of age as confirmed by state identification or passport presented upon completion of the informed consent.
* Participants must have a diagnosis indicative of either Neuropathic or Nociceptive Pain as confirmed with the prescribing medical provider.
* Participants must be starting a new regimen of transdermal (topic) pain therapy with multiple compounded reagents as indicated on prescription from medical provider
* Participants must be willing to participate in the study for a minimum of 12 weeks
* Participants must be able to provide written informed consent.
* Participants must be able to read and understand the english language

Exclusion Criteria:

* Participants must not have prior hypersensitivity or adverse events to any components of the customized prescription as indicated by their allergy history given upon registration at the pharmacy.
* Participants must not be pregnant or planning to become pregnant within the 12 week study period and must not be breastfeeding.
* Participants must not have a diagnosis for cancer in the last 5 years.
* Participants legally authorized representative (LAR) will not be a substitute for the participants' written informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sampling of patients with a diagnosis of neurologic or nociceptive pain whom will be beginning a new regimine of custom compounded pain cream as a pain management therapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Patient Pain Perception | 12 weeks
  Patients will complete surveys every 4 weeks throughout the 12 week evaluation to rate patient pain perception.

SECONDARY OUTCOMES:
Patient overall Sense of Well-Being | 12 weeks
  Patients will complete a survey every 4 weeks throughout the 12 week evaluation to rate their perception of overall well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Akram Z Abu Mahfouz, MS, RPh, Principal Investigator — Marwood Low Cost Pharmacy
Locations (1):
- Marwood Low Cost Pharmacy, Indianapolis, Indiana, United States